CLINICAL TRIAL: NCT01213524
Title: Biological and Behavioral Mechanisms of Smoking in Schizophrenia
Brief Title: Nicotine and Sensorimotor Replacement for Smoking in Smokers With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Tidey, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA014002 (NIH)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-08

CONDITIONS: Tobacco Use Disorder; Schizophrenia
Keywords: nicotine; craving; dual-diagnosis; comorbidity
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Within-subjects design study that investigated the separate and combined effects of sensorimotor replacement for smoking (very low nicotine content [VLNC] cigarettes vs. no cigarettes) and transdermal nicotine replacement (42 mg nicotine [NIC] vs. placebo [PLA] patches). Participants were smokers with schizophrenia and equally-heavy smokers without psychiatric disorders. Each participant underwent the following conditions, in counterbalanced order: VLNC + NIC, VLNC + PLA, no cigarettes + NIC, no cigarettes + PLA, usual-brand cigarettes + no patches.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor were blind to patch condition (NIC or PLA)
Oversight: Data Monitoring Committee: No

ARMS (5):
- Active nicotine replacement (NRT) + denicotinized cigarettes (Active Comparator): 42 mg nicotine replacement plus sensorimotor replacement
  Interventions: Behavioral: sensorimotor replacement; Drug: 42 mg transdermal nicotine replacement
- Placebo NRT + denicotinized cigarettes (Active Comparator): inactive transdermal patches plus sensorimotor replacement
  Interventions: Behavioral: sensorimotor replacement; Drug: Placebo transdermal nicotine
- Active NRT + no cigarettes (Active Comparator): 42 mg nicotine replacement with no sensorimotor replacement
  Interventions: Drug: 42 mg transdermal nicotine replacement
- Placebo NRT + No cigarettes (Placebo Comparator): Double placebo: No nicotine or sensorimotor replacement
  Interventions: Drug: Placebo transdermal nicotine
- usual brand smoking (Active Comparator): positive control: usual brand smoking
  Interventions: Other: usual brand smoking

INTERVENTIONS:
Behavioral: sensorimotor replacement — denicotinized cigarettes
  Arms: Active nicotine replacement (NRT) + denicotinized cigarettes; Placebo NRT + denicotinized cigarettes
Drug: 42 mg transdermal nicotine replacement — 2 21-mg nicotine patches
  Arms: Active NRT + no cigarettes; Active nicotine replacement (NRT) + denicotinized cigarettes
Drug: Placebo transdermal nicotine — 2 placebo patches matched to 21-mg nicotine patches
  Arms: Placebo NRT + No cigarettes; Placebo NRT + denicotinized cigarettes
Other: usual brand smoking — participant smokes usual brand of cigarette
  Arms: usual brand smoking

SUMMARY:
The objective of this study is to investigate the relative contributions of nicotine replacement and sensorimotor replacement (i.e., smoking denicotinized cigarettes) on abstinence-induced smoking urges, withdrawal-related negative affect, psychiatric symptoms, cognitive task performance and 90-min ad libitum usual-brand smoking behavior in smokers with schizophrenia and non-psychiatric smokers.

DETAILED DESCRIPTION:
This study used a mixed between- and within-subjects design to investigate the separate and combined effects of sensorimotor replacement for smoking (very low nicotine content [VLNC] cigarettes vs. no cigarettes) and transdermal nicotine replacement (42 mg nicotine [NIC] vs. placebo [PLA] patches) in smokers with schizophrenia and control smokers without psychiatric illness. Each session contained a 5-h controlled administration period in which participants underwent the following conditions, in counterbalanced order: VLNC + NIC, VLNC + PLA, no cigarettes + NIC, no cigarettes + PLA, Usual Brand cigarettes + no patches. Next, participants completed measures of cigarette craving, nicotine withdrawal, smoking habit withdrawal, cigarette subjective effects, psychiatric symptoms and cognitive task performance followed by a 90-min period of ad libitum usual-brand smoking.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or no psychiatric illness
* 18 and older
* men and women
* cigarette smokers, 20-50 cigarettes per day
* would like to quit someday

Exclusion Criteria:

* medical conditions excluding transdermal nicotine replacement
* pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tidey, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, 121 South Main Street, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community using newspaper and other community advertisements.
Pre-assignment Details: Participants underwent telephone and in-person screening for eligibility.
Groups:
- VLNC + NIC: Within-subjects study with 5 conditions that participants underwent in counter-balanced order:
  1. Transdermal nicotine replacement + sensorimotor replacement (denicotinized cigarettes)
  2. Transdermal nicotine replacement + no sensorimotor replacement
  3. Placebo patches + sensorimotor replacement
  4. Placebo patches + no sensorimotor replacement
  5. Usual brand cigarettes
Period: Baseline
Arm/Group | VLNC + NIC
Started | 75 (Total number who signed informed consent.)
Completed | 68 (Number of participants who continued in the study past baseline)
Not Completed | 7
Not completed — Withdrawal by Subject | 5
Not completed — high breath alcohol levels | 1
Not completed — Physician Decision | 1
Period: Session 2
Arm/Group | VLNC + NIC
Started | 68
Completed | 63 (Number who continued in the study to the next session)
Not Completed | 5
Not completed — Withdrawal by Subject | 5
Period: Session 3
Arm/Group | VLNC + NIC
Started | 63
Completed | 59 (Number who continued in study to next session)
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Session 4
Arm/Group | VLNC + NIC
Started | 59
Completed | 56 (Number who continued in the study to the next session)
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Period: Session 5
Arm/Group | VLNC + NIC
Started | 56
Completed | 56 (Number who continued in the study to the next session)
Not Completed | 0
Period: Session 6
Arm/Group | VLNC + NIC
Started | 56
Completed | 56 (Number who continued in the study to the next session)
Not Completed | 0
Period: Session 7
Arm/Group | VLNC + NIC
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Psychiatric Controls: Smokers without current psychiatric illness
- Total: Total of all reporting groups
Arm/Group | Smokers With Schizophrenia | Non-Psychiatric Controls | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 38 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (8.2) | 41.7 (11.7) | 43.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Preferred Brand Smoke Intake (CO)
Description: preferred brand smoke intake (breath CO) after 5-hr "satiation" periods in which nicotine replacement and sensorimotor replacement were provided under double-blind conditions
Time Frame: 90 min
Population: Participants who completed all conditions and for whom data are available
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- Very Low Nicotine Content Cigarettes + Nicotine Replacement: 5-hr very low nicotine cigarettes + 42 mg nicotine replacement
- Very Low Nicotine Content Cigarettes + Placebo: 5-hr very low nicotine cigarettes + placebo patches
- No Cigarettes + Nicotine Replacement: 5-hr 42 mg nicotine replacement only
- No Cigarettes + Placebo: 5-hr placebo patches only
- Usual Brand Cigarettes: 5-hr use of usual-brand cigarettes
Arm/Group | Very Low Nicotine Content Cigarettes + Nicotine Replacement | Very Low Nicotine Content Cigarettes + Placebo | No Cigarettes + Nicotine Replacement | No Cigarettes + Placebo | Usual Brand Cigarettes
Number analyzed (Participants) | 56 | 56 | 56 | 56 | 56
ppm | 3.30 (8.31) | 3.16 (10.10) | 9.07 (6.95) | 10.54 (7.31) | 5.12 (10.33)

2. Secondary Outcome: Questionnaire on Smoking Urges - Brief Scale (QSU-Brief)
Description: Measure of cigarette craving in which 10 items were rated on 100-mm visual analogue scales (0 = "no urge at all", 100 = "strongest urge you've ever had")
Time Frame: 5 hr
Population: Participants who completed the study and for whom data were available
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Very Low Nicotine Content Cigarettes + Placebo: 5-hr very low nicotine cigarettes plus placebo patches
- Usual Brand Cigarettes: 5-hr use of usual brand cigarettes
Arm/Group | Very Low Nicotine Content Cigarettes + Nicotine Replacement | Very Low Nicotine Content Cigarettes + Placebo | No Cigarettes + Nicotine Replacement | No Cigarettes + Placebo | Usual Brand Cigarettes
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52
mm | 32.02 (32.74) | 37.92 (34.94) | 67.08 (30.33) | 74.13 (26.47) | 24.48 (26.73)

ADVERSE EVENTS:
Arm/Group | Smokers With Schizophrenia | Non-Psychiatric Controls
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 3/37 | 3/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smokers With Schizophrenia (N=37) | Non-Psychiatric Controls (N=38)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — self-report, not related
alcohol detoxification (Nervous system disorders) | 1 (1) | 0 (0) — self-report, not related
suicidality (Psychiatric disorders) | 1 (1) | 0 (0) — self-report, not related
fall requiring stitches (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — self-report, not related
headache (General disorders) | 0 (0) | 1 (1) — self-report, not related
car accident (Social circumstances) | 0 (0) | 1 (1) — self-report, not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes